CLINICAL TRIAL: NCT07213947
Title: Demand and Substitution for Nicotine Pouches Across Dosage
Brief Title: Comparison of Demand and Substitution for Nicotine Pouches as a Function of Nicotine Dosage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Middleton (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, William Middleton, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2372; 5U54DA058256-02 (NIH)
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Tobacco Use; Nicotine Pouch Self-Administration
Keywords: nicotine pouch; behavioral economics; substitution; e-cigarettes; nicotine concentration
MeSH Terms: conditions — Tobacco Use; Vaping

STUDY DESIGN:
Intervention Model Description: Individuals will be asked to purchase nicotine pouches across various prices. Nicotine pouch dosage will be randomly manipulated across pricing conditions. All participants will experience price and dosage changes, but in different orders.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nicotine pouch purchase (Experimental): All participants will be experimentally manipulated by randomizing the dosage of nicotine pouches across varying pricing conditions.
  Interventions: Other: Nicotine Pouch Dosage

INTERVENTIONS:
Other: Nicotine Pouch Dosage — All participants will be experimentally manipulated by having nicotine dosage in hypothetical purchase tasks/ experimental marketplaces altered between market groups.

SUMMARY:
Smoking is a prominent public health issue. Traditional nicotine replacement therapy suffers from being a poor substitute for cigarettes. Novel tobacco products, such as nicotine pouches, show promise as potential low-harm substitutes. Investigators wish to assess the substitutability of cigarettes for nicotine pouches at different dosages and price points. This study will consist of 4000 screened participants online on the crowdsourcing software Prolific, with roughly 400 eligible participants. This study will include the use of an electronic tobacco marketplace.

DETAILED DESCRIPTION:
Participants will be recruited using the crowdsourcing platform Prolific. Prolific has been used by investigators in the past to rapidly recruit a large number of participants. Prolific is powerful due to its ability to sample for specific participant characteristics, such as rurality, while limiting the number of participants who can falsely qualify for the study. This study will screen 4000 tobacco users. Of these we expect to consent 400 nicotine pouch users to the main study. We will then identify their relative rurality through the index of relative rurality.

All potential participants will complete a series of demographic questions related to tobacco use, exposure to tobacco marketing, behavioral factors, and rurality, which will act as predictors of susceptibility to nicotine pouch initiation. All participants' Zip-code will be sampled and transformed into Index of Relative Rurality scores to assess rurality continuously. Data for nicotine pouch users will be assessed using multivariable regression-based analysis with interactions to determine which factors influence susceptibility to products other than nicotine pouches, and the effect of index of relative rurality on the relationship between predictors and initiation. Nicotine pouch users will continue on to an experimental tobacco marketplace (ETM) that will assess their valuation of nicotine pouches against other tobacco products, which will serve as a proxy to their likelihood to switch from nicotine pouches when the cost required to obtain nicotine pouches increases. Participants will complete 8 scenarios with escalating prices for nicotine pouches. Participants will be exposed to a virtual store and prompted to purchase as many tobacco products as they wish with an unlimited budget for their weekly supply of tobacco products. After making a set of purchases, participants will continue on to a subsequent marketplace where the price of their preferred product is increased. The degree to which participants purchase other tobacco products as nicotine pouch price increases will constitute demand. Demand will be analyzed using multilevel modeling methods to produce relevant demand indices. Participants will then have to complete 5 marketplaces of 8 price conditions. In each marketplace, the nicotine dosage of nicotine pouches will be randomly assigned to either 0 milligrams, 2 milligrams, 4 milligrams, 6 milligrams, or 8 milligrams.

ELIGIBILITY:
Inclusion Criteria:

* tobacco users will be eligible for a general screener
* nicotine pouch users will be eligible for the full marketplace study
* users of the crowdsourcing website Prolific

Exclusion Criteria:

* non nicotine pouch user
* <18+ years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1360 (Actual)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-01-02 (Actual); Study Completion 2026-01-02 (Actual)

PRIMARY OUTCOMES:
Nicotine Pouch Demand Indices | Within 1 hour of enrollment, participants are expected to have completed the full trial.
  Behavioral demand curves will be drawn for nicotine pouch consumption as a function of price. Demand curves will be compared across dosage conditions on three indices: breakpoint (price at which consumption drops to zero) , elasticity of demand (rate of decline of consumption at any price), and intensity of demand (consumption at zero price).

SECONDARY OUTCOMES:
Substitution of Nicotine Pouches for other Tobacco Products | Within 1 hour of enrollment participants are expected to have completed the whole trial.
  The experimental tobacco marketplace will also include a variety of other tobacco products. Investigators will examine whether individuals begin consuming other products as the price of nicotine pouches increases. Examining substitution for combustible and e-cigarettes is a secondary outcome.
Effects of Relative Rurality on Nicotine Pouch Demand and Substitution | Within 1 hour of enrollment participants are expected to have completed the whole trial.
  The Index of Relative Rurality will be used to compare demand for nicotine pouches across dosages and substitution effects across an all encompassing spectrum of rurality to determine whether urbanity, periurbanity, or rurality are risk profiles for harmful tobacco consumption

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Koffarnus, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Turfland Medical Center, Department of Family and Community Medicine, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT07213947/ICF_000.pdf